CLINICAL TRIAL: NCT07078968
Title: A REAL WORLD DATA COLLECTION OF HUMAN AMNIOTIC MEMBRANE(S) ON DIABETIC FOOT ULCERS, VENOUS LEG ULCERS, PRESSURE ULCERS AND POST OPERATIVE WOUNDS
Status: Active, not recruiting | Type: Observational
Sponsor: BioLab Holdings (Industry)
Responsible Party: Sponsor
Other Study IDs: RWE-001-25
Record Dates: First submitted 2025-07-14; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Venous Leg Ulcer (VLU); Diabetic Foot Ulcer (DFU); Pressure Ulcer (PU)
MeSH Terms: conditions — Varicose Ulcer; Diabetic Foot; Pressure Ulcer | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Group 1 Amniotic Membrane: De-Identified subject data will be extracted from investigators' medical records for subjects who received Tri-Membrane Wrap™, Membrane Wrap™, Membrane Wrap-Hydro™ plus SOC in subjects with eligible DFUs, VLUs, PUs and post operative wounds
  Interventions: Device: Tri-Membrane Wrap™; Device: Membrane Wrap™; Device: Membrane Wrap-Hydro™
- Group 2 SOC: De-identified subject data will be extracted from investigators' medical records who were treated with only Standard of Care with eligible DFUs, VLUs, PUs and post operative wounds. Subjects in the SOC may have received hyperbaric or wound vac therapies as part of their treatments.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Device: Tri-Membrane Wrap™ — Membrane Wrap™
  Groups: Group 1 Amniotic Membrane
Device: Membrane Wrap™ — Membrane Wrap™
  Groups: Group 1 Amniotic Membrane
Device: Membrane Wrap-Hydro™ — Membrane Wrap-Hydro™
  Groups: Group 1 Amniotic Membrane
Other: Standard of Care — Basic care involves debridement, along with local wound care depending on the wound needs. Debridement involves removal of fibrin and devitalized tissue from the base and the borders of the ulcer which is necessary in all treatment plans to reduce the risk of infection and promote healing.
  Groups: Group 2 SOC

SUMMARY:
This study is designed to evaluate the effectiveness of Tri-Membrane Wrap™, Membrane Wrap™ and Membrane Wrap-Hydro™ compared to the effectiveness of Standard of Care alone though a retrospective data collection.

DETAILED DESCRIPTION:
This is a retrospective multi-center study collecting real world evidence on the use of Tri-Membrane Wrap™, Membrane Wrap™, Membrane Wrap-Hydro™ and Standard of Care alone in subjects with eligible DFUs, VLUs, PUs, and post operative wounds that have not healed with conventional therapy for greater than or equal to 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Subject had the presence of diabetic foot ulcers, Venous insufficiency ulcers, pressure ulcers and/or post-operative wounds
2. Subject has retrospectively been treated with Tri-Membrane Wrap™, Membrane Wrap™ and Membrane Wrap-Hydro™ or Subject has retrospectively been treated with Standard of Care only.
3. Subjects should have been treated from January 2022 to present day.

Exclusion Criteria:

1. Subjects that did not have a wound closure verification appointment.
2. Any subject who received any product other than Tri-Membrane Wrap™, Membrane Wrap™ and Membrane Wrap-Hydro™ during their treatment time.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with difficult to heal partial- or full-thickness diabetic foot ulcers (DFU), venous leg ulcers (VLU), pressure ulcers (PU), and post-operative wounds defined as an ulcer that has not healed with conventional therapy for ≥ 4 weeks.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-04-23 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Frequency of wound closure by or on week 16 | 16 weeks
  Wound closure is defined as: Full epithelialization of the wound with the absence of drainage. Epithelialization is defined as a layer of epithelium visible on the wound surface

SECONDARY OUTCOMES:
Wound improvement by or on End of Study (EOS) from baseline | 16 weeks
  Defined by: >60% reduction in area, or >60% reduction in depth, or >75% reduction in volume
Incidence of wound recurrence within the 16-week study period | 16 weeks
  Incidence of wound recurrence within the 16-week study period
Mean number of wound free days within the 16-week study period | 16 weeks
  Mean number of wound free days within the 16-week study period

CONTACTS AND LOCATIONS:
Overall Officials: Marshall Medley, Study Chair — Sponsor GmbH
Locations (4):
- United States (4):
  - Athena Specialty Group, Phoenix, Arizona
  - Revive Advanced Wound Care, Toms River, New Jersey
  - Houston Foot and Ankle Care, Houston, Texas
  - Houston Foot Dr, Houston, Texas

IPD SHARING:
Plan to Share IPD: No